CLINICAL TRIAL: NCT03885505
Title: An Analysis of the Quality of Life and Sexual Quality of Life of Cervical Cancer Radiotherapy Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, HONGNAN ZHEN, department of radiation oncology, Peking Union Medical College Hospital
Other Study IDs: ZHN 20181125
Record Dates: First submitted 2018-11-25; First posted 2019-03-21 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Cervical Cancer; Radiotherapy Side Effect; Quality of Life
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cervical cancer radiotherapy patients have a decline in quality of life and sexual quality of life

DETAILED DESCRIPTION:
Objective: To investigate the quality of life and sexual quality of life and its influencing factors in cervical cancer undergoing radiotherapy patients.

Methods:The cervical cancer cancer scale (FACT-Cx4.0) and the female sexual function index (FSFI) in the cancer treatment function evaluation system were used. The quality of life and sexual quality of life of cervical cancer patients undergoing radiotherapy in PUMC Hospital were analyzed and scored to analyze the effects of age, education level, clinical stage and treatment methods on the quality of life and sexual quality of life of cervical cancer radiotherapy patients

ELIGIBILITY:
Inclusion Criteria:

* adult female
* diagnosed with cervical cancer' and acquire therapy as part of treatment
* undertaken or have finished radiotherapy in Peking Union Medical College Hospital
* agreed with informed consent

Exclusion Criteria:

* with cognitive dysfunction or cannot fulfilled the questionaire
* refuse or quit the research
* submit questionnaire with missing information

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical cancer patients treated by radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-25 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
using fact-cx4.0 to evaluate the qol of cervical cancer patients undergoing radiotherapy | through study completion, an average of half a year
  Functional Assessment of Cancer Therapy-Cervix V4.0 (FACT-Cx V4.0) was used to evaluate patients'quality of life. The scale is composed of general cancer quality of life assessment scale (FACT-G) and cervical cancer specific module (CCS). It contains 5 dimensions and 42 subjects. The higher the score of positive questions, the better the quality of life. The higher the score of reverse questions, the worse the quality of life. If it is a reverse question, the original score of this question is subtracted by 4. The higher the total score, the better the quality of life. The study was conducted by face-to-face investigation of specialist nurses. All patients'investigation data were kept strictly confidential.
  And follow the principles of medical ethics.using spss to analysis the data.

SECONDARY OUTCOMES:
using fsfi to evaluate the qol of cervical cancer patients undergoing radiotherapy | through study completion, an average of half a year
  Female Sexual Function Index (FSFI) was used to measure the quality of sexual life. The higher the score of positive items, the worse the quality of sexual life. If the reverse items were negative, the original score of the item could be subtracted by 5. The higher the total score, the better the quality of sexual life. The study was conducted by face-to-face investigation by specialist nurses. All patients'investigation data were strictly confidential and followed the medical ethics principles.using spss to analysis the data.

IPD SHARING:
Plan to Share IPD: Undecided